CLINICAL TRIAL: NCT06433102
Title: Assessing the Effectiveness of Visual Perception Training Based on Lateral Masking Paradigm in Glaucoma Patients
Brief Title: Evaluation of Visual Training System in Patients With Glaucoma
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023KYPJ008
Record Dates: First submitted 2024-05-22; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-02

CONDITIONS: Glaucoma
Keywords: Visual perceptual training; Vision rehabilitation; Glaucoma; Lateral masking paradigm
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: The technical staff and research assistants involved in subject enrollment, outcome measurement, and data collection are blinded to the intervention allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the training group (Experimental): Participants in this group received visual perceptual training based on the lateral masking paradigm every other day for 35 to 45 minutes, with each cycle consisting of 40 sessions, lasting approximately 3 months. The training began in the hospital during the first week and continued at home using personal computers thereafter. The personal computers were connected to a central server via the internet.
  Interventions: Other: Visual perceptual training based on the lateral masking paradigm
- the control group (No Intervention): The control group maintained the original treatment plan without any additional interventions.

INTERVENTIONS:
Other: Visual perceptual training based on the lateral masking paradigm — Visual perceptual training is a novel rehabilitation approach aimed at enhancing visual performance through practice of visual tasks. Patients received visual perceptual training based on the lateral masking paradigm every other day. Each training session consisted of 9 stages, totaling 900 trials, lasting 35 to 45 minutes. The stimuli consisted of a central Gabor patch with relatively low contrast positioned in the central fixation area, along with co-linear high-contrast Gabor patches distributed above and below the central stimulus. These stimuli were presented on a Liquid Crystal Display (LCD) monitor, with a training distance of 150 cm.
  Arms: the training group

SUMMARY:
This study intends to conduct visual function examinations and follow-ups on two groups of glaucoma patients, one receiving visual perceptual training and the other serving as a control without training. The aim of this study is to explore the effects of visual perceptual training based on the lateral masking paradigm on patients' visual function. Additionally, synchronized EEG-fNIRS signals will be collected to investigate whether changes in patients' visual function are accompanied by corresponding alterations in brain function.

DETAILED DESCRIPTION:
Glaucoma is a chronic eye disease that causes irreversible damage to the optic nerve and can lead to severe vision loss and blindness. In China, the blindness rate among glaucoma patients is 22.7%, accounting for 8.8% of the total blind population. Among individuals aged 40 and above in urban and rural areas of China, approximately 9.2 million suffer from glaucoma, with 55% experiencing blindness in at least one eye and 18.1% experiencing blindness in both eyes [1,2]. Glaucoma patients may experience severe impairment in visual function, leading to significant limitations in vision-related activities such as mobility and visual searching. This has a negative impact on the quality of life (QOL) of patients, increasing the burden on individuals, families, and society.

Vision Rehabilitation (VR) is an integral component of the eye care continuum, spanning from diagnosis to treatment and rehabilitation [3]. It aims to assist visually impaired patients in maximizing their remaining vision, facilitating easier performance of daily activities, promoting independence, and enhancing quality of life (QOL). However, for glaucoma patients with visual field defects, traditional methods such as inverted telescopes and prism glasses are plagued by shortcomings such as unattractive appearance, bulkiness, blurred visual quality, and challenges in adaptation.

Perceptual Learning (PL) is a novel rehabilitation approach aimed at enhancing visual performance through intensified practice of visual tasks. Many studies have shown that visual perceptual training can improve visual function in patients with different types of amblyopia or presbyopia, as the nervous system exhibits significant neuroplasticity [4-6]. However, there is limited research on visual perceptual training in visual rehabilitation for glaucoma.

Therefore, this study intends to conduct visual function examinations and follow-ups on two groups of glaucoma patients, one receiving visual perceptual training and the other serving as a control without training. The aim of this study is to explore the effects of visual perceptual training based on the lateral masking paradigm on patients' visual function. Additionally, synchronized EEG-fNIRS signals will be collected to investigate whether changes in patients' visual function are accompanied by corresponding alterations in brain function.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 10 years old
2. diagnosed with primary glaucoma or developmental glaucoma
3. the best corrected visual acuity ≥0.1 and the mean deviation of the visual field worse or equal to -6 dB
4. visual acuity, intraocular pressure, and other eye conditions have been stable for more than 3 months
5. participants capable of understanding the purpose of the study and providing informed consent
6. participants capable of cooperating with relevant examinations.

Exclusion Criteria:

1. a history of eye surgery or eye laser within three months
2. complicated with other ophthalmopathy affecting visual function (except cataract, ametropia), such as age-related macular degeneration, diabetic retinopathy, optic nerve disease, retinal vascular disease, etc.
3. serious systemic diseases, such as neurological diseases, cardiovascular diseases, psychological diseases, malignant tumors, etc
4. pregnant or lactating women.

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-06-03 (Estimated); Primary Completion 2025-04-26 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Contrast sensitivity function | 6 months after intervention
  Contrast sensitivity function (CSF) was assessed using the qCSF method at baseline, and at 1 day, 3 months, and 6 months after the intervention. The qCSF method employed a Bayesian adaptive learning procedure. Data collected for analysis included contrast sensitivity at 19 spatial frequencies, the area under the log CSF (AULCSF), and the cutoff spatial frequency.

SECONDARY OUTCOMES:
Visual field | 6 months after intervention
  Visual field testing was conducted using automated perimetry with the 30-2 Swedish interactive threshold algorithm. The examination was performed at baseline and 1 day, 3 months, and 6 months after the intervention.
Visual acuity | 6 months after intervention
  Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity chart was used. The examination was performed at baseline and 1 day, 3 months, and 6 months after the intervention.
Stereoacuity | 6 months after intervention
  Stereoacuity was measured using the Titmus stereopsis test at baseline, as well as 1 day, 3 months, and 6 months after the intervention.
Glaucoma Visual Functioning Questionnaire-40 (GVFQ-40) | 6 months after intervention
  The GVFQ-40 consists of 40 items and measures the difficulty of daily activities of glaucoma patients in five domains of functioning (mobility, visual tracking, reading, identification and night vision ). Each item has six answer options, that is, no difficulty (score = 1), mild difficulty (score = 2), moderate difficulty (score = 3), extremely difficult (score = 4), completely unable to complete (score = 5), and do not perform for nonvisual reasons (no score). The GVFQ-40 was administered at baseline and 1 day, 3 months, and 6 months after the intervention.
National Eye Institute-Visual Function Questionnaire-25 (NEI VFQ-25) | 6 months after intervention
  The National Eye Institute-Visual Function Questionnaire-25 (NEI VFQ-25) is a valid and reliable vision-related quality of life (QOL) questionnaire designed for persons who have chronic eye diseases or low vision. It includes 25 items that comprise 11 subscales on different aspects of vision-related functioning and QOL and 1 item on general health. NEI VFQ-25 scores range from 0 to 100, with a higher score representing better functioning. The NEI VFQ-25 was administered at baseline and 1 day, 3 months, and 6 months after the intervention.
Reach-and-Grasp Kinematics | 6 months after intervention
  The reaching-and-grasping (prehension) task was conducted to assess patients' eye-hand coordination abilities at baseline and 1 day, 3 months, and 6 months post-intervention. The motion capture system recorded the movements of the preferred hand. Various metrics of prehension planning and online control were measured, including initiation time, total movement duration, peak velocity, and other relevant parameters.
Electroencephalogram (EEG) node efficiency | 6 months after intervention
  Electroencephalogram was performed to track the electrical activity of the brain in real time at baseline and 1 day, 3 months, and 6 months after the intervention. Node efficiency was calculated. Node efficiency is a metric that characterizes the efficiency of a single node in connecting with all other parts of the network. It reflects the centrality and importance of a node within the network.
Functional near-infrared spectroscopy (fNIRS) | 6 months after intervention
  Functional near-infrared spectroscopy (fNIRS) was conducted to capture spatial information on cerebral blood flow and oxygenation conditions at baseline, as well as 1 day, 3 months, and 6 months after the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Opthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Foster PJ, Johnson GJ. Glaucoma in China: how big is the problem? Br J Ophthalmol. 2001 Nov;85(11):1277-82. doi: 10.1136/bjo.85.11.1277. PMID 11673287
- [Background] Fontenot JL, Bona MD, Kaleem MA, McLaughlin WM Jr, Morse AR, Schwartz TL, Shepherd JD, Jackson ML; American Academy of Ophthalmology Preferred Practice Pattern Vision Rehabilitation Committee. Vision Rehabilitation Preferred Practice Pattern(R). Ophthalmology. 2018 Jan;125(1):P228-P278. doi: 10.1016/j.ophtha.2017.09.030. Epub 2017 Nov 4. No abstract available. PMID 29108747
- [Background] Matteo BM, Vigano B, Cerri CG, Perin C. Visual field restorative rehabilitation after brain injury. J Vis. 2016 Jul 1;16(9):11. doi: 10.1167/16.9.11. PMID 27472498
- [Background] Polat U, Ma-Naim T, Belkin M, Sagi D. Improving vision in adult amblyopia by perceptual learning. Proc Natl Acad Sci U S A. 2004 Apr 27;101(17):6692-7. doi: 10.1073/pnas.0401200101. Epub 2004 Apr 19. PMID 15096608
- [Background] Zhong J, Wang W, Li J, Wang Y, Hu X, Feng L, Ye Q, Luo Y, Zhu Z, Li J, Yuan J. Effects of Perceptual Learning on Deprivation Amblyopia in Children with Limbal Dermoid: A Randomized Controlled Trial. J Clin Med. 2022 Mar 28;11(7):1879. doi: 10.3390/jcm11071879. PMID 35407483